CLINICAL TRIAL: NCT05111301
Title: Control-IQ Technology in Individuals With Type 2 Diabetes (2IQ)
Brief Title: Control-IQ Technology in Individuals With Type 2 Diabetes
Acronym: 2IQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0009569
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: type 2 diabetes; Control-IQ technology; automated insulin dosing; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Basal Insulin Only (Group A) (Experimental): * 2 to 4 week CGM run-in
  * 2 to 4 week pump run-in
  * 6 weeks Control-IQ technology use
  Interventions: Device: Control-IQ technology 1.5
- Multiple Daily Injections (Group B) (Experimental): * 2 to 4 week CGM run-in
  * 2 to 4 week pump run-in
  * 6 weeks Control-IQ technology use
  Interventions: Device: Control-IQ technology 1.5

INTERVENTIONS:
Device: Control-IQ technology 1.5 — All subjects wearing the t-slim X2 insulin pump with Control-IQ technology 1.5, and wearing the Dexcom G6 sensor.
  Outcomes will be analyzed overall and subgroup analysis will be performed by Group, and by baseline A1c level.

SUMMARY:
A prospective, multicenter study of 6 weeks of home use of Control-IQ technology in individuals with type 2 diabetes age 18 and older.

DETAILED DESCRIPTION:
The objective of this prospective, multicenter study is to assess safety and explore glycemic outcomes associated with use of Control-IQ technology in adults with type 2 diabetes who require insulin. After an initial run-in period, all participants will use the study system (pump and CGM) for 6 weeks. Participants will perform exercise challenges once each week during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and residing in the US
* Clinical diagnosis, based on investigator assessment, of type 2 diabetes for at least one year
* Using a stable insulin dose for at least 3 months, to include A) basal insulin only, or B) MDI, to include CSII (including use of AID systems other than Tandem Control-IQ technology)
* Total daily insulin dose ≤200 units/day
* Willing to use only aspart (novolog) or lispro (humalog) insulin with the study pump, with no use of concentrated insulin above U-100, long-acting basal insulin injections, or inhaled insulin
* For females, not currently known to be pregnant
* If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* HbA1c ≥ 7.5% and ≤ 12% at screening
* Has current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (will provide prescription if they do not have one)
* Be willing to exercise for 30 minutes or more at least once per week during the main phase of the study
* Has the ability to read and understand written English
* Investigator believes that the participant can successfully and safely operate all study devices and is capable of adhering to the protocol and completing the study.

Exclusion Criteria:

* Prior use of Tandem t:slim X2 insulin pump with Control-IQ technology
* Two or more episodes of severe hypoglycemia (needing assistance) in the past 6 months
* History of inpatient psychiatric treatment in the past 6 months
* History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or unwillingness to agree to abstain from illicit drugs throughout the study.
* History of significant heart disease, lung disease, liver disease, chronic kidney disease, or other systemic disease determined by investigator to interfere with the study, or make required exercise unsafe
* History of significant vision, hearing, or dexterity problems that will impair use of the closed loop system
* Use of glucocorticoids, beta blockers, sulfonylureas, meglitinides or other medications specifically listed in the protocol or determined by investigator to interfere with the study
* Unstable dose of SGLT-2 inhibitor, GLP-1 receptor agonist, or other adjuvant medication specifically listed in the protocol, or starting a new glucose lowering agent during the trial.
* Unstable dose of any medication used for weight loss, as listed in the protocol, or starting a new medication for weight loss during the trial.
* Abnormal screening electrocardiogram consistent with increased risk during exercise, such as arrhythmia, ischemia, or prolonged QTc interval (>450 ms)
* History of hemodialysis
* History of adrenal insufficiency
* Uncontrolled hypo- or hyperthyroidism
* Significant diabetes related complications, based on investigator assessment
* Immediate family member (spouse, biological or legal guardian, child, sibling, parent) who is an investigative site personnel directly affiliated with this study or who is an employee of Tandem Diabetes Care, Inc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Levy, MD, Study Chair — Icahn School of Medicine at Mt. Sinai
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Texas Diabetes and Endocrinology, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levy CJ, Raghinaru D, Kudva YC, Pandit K, Blevins T, Casaubon L, Desjardins D, Levister CM, O'Malley G, Reid C, Lum J, Kollman C, Beck RW. Beneficial Effects of Control-IQ Automated Insulin Delivery in Basal-Bolus and Basal-Only Insulin Users With Type 2 Diabetes. Clin Diabetes. 2024 Winter;42(1):116-124. doi: 10.2337/cd23-0025. Epub 2023 Aug 28. PMID 38230336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 3 clinical centers in the United States. All eligible participants were included without regard to gender, race, or ethnicity. Each site was asked to contribute ~10 participants (5 basal only / 5 MDI) toward the overall recruitment goal.
Groups:
- Basal Insulin Only (Group A); Multiple Daily Injections (Group B): * 2 to 4 week CGM run-in
  * 2 to 4 week pump run-in
  * 6 weeks Control-IQ technology use
  Control-IQ technology 1.5: All subjects wearing the t-slim X2 insulin pump with Control-IQ technology 1.5, and wearing the Dexcom G6 sensor.
  Outcomes will be analyzed overall and subgroup analysis will be performed by Group, and by baseline A1c level.
Period: Overall Study
Arm/Group | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Started | 13 | 17
Completed | 13 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B) | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12) | 54 (12) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 9 | 14 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent of glycated hemoglobin] | 8.2 (0.9) | 8.9 (1.3) | 8.6 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: CGM Time Below 54 mg/dL
Description: CGM-measured percentage below 54 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- Overall; Basal Insulin Only (Group A); Multiple Daily Injections (Group B): * 2 to 4 week CGM run-in with insulin injections (baseline)
  * 2 to 4 week open loop with insulin pump and Dexcom G6 sensor
  * 6 weeks Control-IQ technology 1.5 use
  Control-IQ technology 1.5: All subjects wearing the t:slim X2 insulin pump with Control-IQ technology 1.5, and wearing the Dexcom G6 sensor.
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.00]
  Open-Loop | 0.00 [0.00 to 0.08] | 0.00 [0.00 to 0.12] | 0.00 [0.00 to 0.03]
  Control-IQ | 0.02 [0.00 to 0.07] | 0.02 [0.01 to 0.08] | 0.02 [0.00 to 0.05]

2. Primary Outcome: CGM Time Above 180 mg/dL
Description: CGM-measured percentage above 180 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 44 (25) | 39 (15) | 48 (31)
  Open-Loop | 37 (20) | 34 (22) | 39 (19)
  Control-IQ | 29 (18) | 26 (15) | 31 (20)
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.004, t-test, 2 sided

3. Secondary Outcome: CGM Time In Range 70-180 mg/dL
Description: CGM-measured percentage in range 70-180 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 56 (25) | 61 (15) | 52 (31)
  Open-Loop | 63 (20) | 66 (22) | 61 (18)
  Control-IQ | 71 (18) | 74 (15) | 68 (20)
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.004, t-test, 2 sided

4. Secondary Outcome: CGM Time Below 70 mg/dL
Description: CGM-measured percentage below 70 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 0.05 [0.00 to 0.47] | 0.00 [0.00 to 0.25] | 0.11 [0.00 to 0.47]
  Open-Loop | 0.10 [0.00 to 0.51] | 0.19 [0.00 to 0.35] | 0.03 [0.00 to 0.60]
  Control-IQ | 0.12 [0.04 to 0.34] | 0.09 [0.05 to 0.25] | 0.13 [0.03 to 0.36]
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.54, t-test, 2 sided

5. Secondary Outcome: CGM Time Above 250 mg/dL
Description: CGM-measured percentage above 250 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 8.5 [1.7 to 21.1] | 12.9 [1.7 to 14.7] | 6.8 [2.4 to 29.6]
  Open-Loop | 6.7 [2.1 to 12.2] | 8.1 [0.9 to 16.9] | 6.3 [3.8 to 10.0]
  Control-IQ | 2.9 [1.1 to 12.8] | 1.9 [0.8 to 7.5] | 2.9 [1.3 to 13.1]
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.03, t-test, 2 sided

6. Secondary Outcome: CGM Time In Range 70-140 mg/dL
Description: CGM-measured percentage in range 70-140 mg/dl, compared to baseline
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of time
  Baseline | 30 (17) | 32 (13) | 28 (20)
  Open-Loop | 34 (22) | 38 (23) | 31 (21)
  Control-IQ | 42 (18) | 45 (17) | 40 (19)
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.001, t-test, 2 sided

7. Secondary Outcome: CGM Mean Glucose mg/dL
Description: CGM measured mean glucose mg/dL, compared to baseline
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
mg/dL
  Baseline | 184 (42) | 174 (22) | 192 (52)
  Open-Loop | 172 (32) | 170 (35) | 174 (30)
  Control-IQ | 163 (28) | 159 (23) | 166 (32)
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.01, t-test, 2 sided

8. Secondary Outcome: Coefficient of Variation (CV)
Description: CGM measured glucose variability measured with the coefficient of variation (CV), compared to baseline
Time Frame: 14 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of coefficient of variation
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
percentage of coefficient of variation
  Baseline | 28 [24 to 31] | 29 [27 to 31] | 25 [23 to 32]
  Open-Loop | 29 [23 to 34] | 30 [23 to 31] | 29 [23 to 34]
  Control-IQ | 28 [24 to 31] | 27 [24 to 30] | 30 [24 to 31]
Statistical Analysis 1: Comparison: Overall; For Control-IQ Versus Baseline; Test type: Superiority; p = 0.80, t-test, 2 sided

9. Other Pre Specified Outcome: Severe Hypoglycemia (Needing Assistance)
Description: The number of severe hypoglycemic events (needing assistance)
Time Frame: 14 weeks
Measure: Number; unit: events
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
events | 0 | 0 | 0

10. Other Pre Specified Outcome: DKA
Description: The number of DKA events
Time Frame: 14 weeks
Measure: Number; unit: events
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
events | 0 | 0 | 0

11. Other Pre Specified Outcome: Hyperosmolar Hyperglycemic Syndrome
Description: The number of Hyperosmolar Hyperglycemic Syndrome events
Time Frame: 14 weeks
Measure: Number; unit: events
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
events | 0 | 0 | 0

12. Other Pre Specified Outcome: All Serious Adverse Events
Description: The number of Serious Adverse Events
Time Frame: 14 weeks
Measure: Number; unit: events
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
events | 0 | 0 | 0

13. Other Pre Specified Outcome: Unanticipated Adverse Device Effects
Description: The number of Unanticipated Adverse Device Effects
Time Frame: 14 weeks
Measure: Number; unit: events
Arm/Group | Overall | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
Number analyzed (Participants) | 30 | 13 | 17
events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Basal Insulin Only (Group A) | Multiple Daily Injections (Group B)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 1/13 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Insulin Only (Group A) (N=13) | Multiple Daily Injections (Group B) (N=17)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) — During CGM-Run Period
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Due To Infusion Set Failure
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Related To Illness
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT05111301/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05111301/SAP_001.pdf